CLINICAL TRIAL: NCT02047370
Title: Effects of Manual Therapy in Patients With Asthma
Brief Title: Manual Therapy in Patients With Asthma
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The sample size was not completed
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0046UG
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: stretching, diaphragm, asthma, manual therapy
MeSH Terms: conditions — Asthma | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diaphragm stretching (Experimental): 30 Patients with asthma are included in this group. They will receive a diaphragm stretching technique
  Interventions: Other: Diaphragm stretching
- Placebo group (Placebo Comparator): Ultrasound disconnected in same position and with the same duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Diaphragm stretching — The therapist stands behind the patient and passes his hands around the thoracic cage, carefully introducing fingers under the costal margins. The patient slightly rounds the trunk in order to relax rectus abdominis. During the exhalation of the patient the therapist grasps the lower ribs and costal margin and eases the hands caudally. This traction was maintained during 5-7 minutes.
  Other Names: Manual therapy
  Arms: Diaphragm stretching
Other: Placebo — The same therapist, patient position and duration of the technique, but using disconnected ultrasound
  Other Names: Disconnected ultrasound.
  Arms: Placebo group

SUMMARY:
Physical therapists have traditionally included various forms of manual therapy among the therapeutic approaches to respiratory conditions. The aim of this study was to evaluate the effect of diaphragmatic stretching technique on pulmonary ventilation, rig bage excursion and spirometric values in patients diagnosed with asthma.

DETAILED DESCRIPTION:
Asthma is a chronic lung disease involving an inflammation and a narrowing of the airways. Asthma causes wheezing, chest tightness, shortness of breath, and coughing.

A variety of manual therapies are commonly used to treat patients with asthma. There is a need to conduct studies in order to examine the effects of manual therapies on clinically relevant outcomes. Techniques aim to increase movement in the rib cage and the spine to try and improve the working of the lungs and circulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 18 and 45 years.
* Diagnosis of asthma.
* No exacerbations during last month.

Exclusion Criteria:

* History of spine surgery.
* Diabetes, neurological or a cardiovascular disease.
* Spine deformities and use of orthopedic devices.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity | Baseline, 7 days
  The amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. It is going to be measured using a spirometer as recommended by the American Thoracic Society.

SECONDARY OUTCOMES:
Abdominal Kinematics | baseline, 7 days
  Abdominal kinematic measurements can be used as an evaluative method to quantify possible alterations in abdominal movements.
Airway diffusing capacity | baseline, 7 days
  The airway diffusion capacity will be measure using the deep breeze device. This is a non-invasive and radiation-free gadget that provides a dynamic image of the lungs, delivering both structural and functional information.
Forced expiratory volume in the first second | baseline, 7 days
  This is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. It is going to be measured using a spirometer as recommended by the American Thoracic Society.
Rib cage excursion | baseline, 7 days
  Rib cage excursion can be used as an evaluative method for diaphragmatic breathing excursion to quantify possible alterations in thoracic capacity and chest wall compliance as achieved by all expiratory and inspiratory muscles

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of health Sciences. University of Granada, Granada, Spain, Spain